CLINICAL TRIAL: NCT06868667
Title: DREAMM 7: A Multicenter, Open-Label, Randomized Phase III Study to Evaluate the Efficacy and Safety of the Combination of Belantamab Mafodotin, Bortezomib, and Dexamethasone (B-Vd) Compared With the Combination of Daratumumab, Bortezomib and Dexamethasone (D-Vd) in Participants With Relapsed/Refractory Multiple Myeloma
Brief Title: Japan Expansion Cohort: Evaluation of Efficacy and Safety of Belantamab Mafodotin, Bortezomib and Dexamethasone Versus Daratumumab, Bortezomib and Dexamethasone in Participants With Relapsed/Refractory Multiple Myeloma
Acronym: DREAMM 7
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207503-JPN
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Japan Expansion Cohort; Belantamab mafodotin; Relapsed/refractory multiple myeloma; Daratumumab; Bortezomib; Dexamethasone; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Belantamab mafodotin and Bortezomib plus Dexamethasone (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Bortezomib; Drug: Dexamethasone
- Daratumumab and Bortezomib plus Dexamethasone (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab mafodotin — Humanized anti-B-cell maturation antigen (BCMA) antibody/drug conjugate.
  Arms: Belantamab mafodotin and Bortezomib plus Dexamethasone
Drug: Daratumumab — Anti-cluster of differentiation 38 [CD-38] monoclonal antibody.
  Arms: Daratumumab and Bortezomib plus Dexamethasone
Drug: Bortezomib — Proteasome Inhibitor.
Drug: Dexamethasone — Synthetic glucocorticoid with anti-tumor activity.

SUMMARY:
This study is designed to evaluate safety and efficacy of belantamab mafodotin in combination with bortezomib/dexamethasone versus daratumumab in combination with bortezomib/dexamethasone in the Japanese participants with relapsed refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma as defined by the International Myeloma Working Group (IMWG) criteria.
* Previously treated with at least 1 prior line of multiple myeloma (MM) therapy and must have documented disease progression during or after their most recent therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Must have at least 1 aspect of measurable disease, defined as one of the following;

  1. Urine M-protein excretion >=200 mg per 24-hour, or
  2. Serum M-protein concentration >=0.5 grams per deciliter (g/dL), or
  3. Serum free light chain (FLC) assay: involved FLC level >=10 mg per dL (>=100 mg per liter) and an abnormal serum free light chain ratio (<0.26 or >1.65).
* All prior treatment-related toxicities (defined by National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI-CTCAE] version 5.0) must be <=Grade 1 at the time of enrollment, except for alopecia.
* Adequate organ function

Exclusion Criteria:

* Intolerant to daratumumab.
* Refractory to daratumumab or any other anti-CD38 therapy (defined as progressive disease during treatment with anti-CD38 therapy, or within 60 days of completing that treatment).
* Intolerant to bortezomib, or refractory to bortezomib (defined as progressive disease during treatment with a bortezomib-containing regimen of 1.3 mg/m^2 twice weekly, or within 60 days of completing that treatment). Note: participants with progressive disease during treatment with a weekly bortezomib regimen are allowed.
* Ongoing Grade 2 or higher peripheral neuropathy or neuropathic pain.
* Prior treatment with anti-B-cell maturation antigen (anti-BCMA) therapy.
* Prior allogenic stem cell transplant.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions, including renal, liver, cardiovascular, or certain prior malignancies.
* Corneal epithelial disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2026-06-19 (Estimated)

CONTACTS AND LOCATIONS:
Locations (16):
- Japan (16):
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Himeji
  - GSK Investigational Site, Kamakura
  - GSK Investigational Site, Kitakyushu
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Matsuyama
  - GSK Investigational Site, Nagoya
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōgaki
  - GSK Investigational Site, Shibukawa
  - GSK Investigational Site, Sunto-gun
  - GSK Investigational Site, Suwa
  - GSK Investigational Site, Toyohashi
  - GSK Investigational Site, Yokohama

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Groups:
- Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex): Japanese participants with Relapsed/Refractory Multiple Myeloma (RRMM) received intravenous (IV) infusion of 2.5 milligram (mg)/kilogram (kg) belantamab mafodotin on Day 1 of each 21-day Cycle until disease progression, intolerable toxicity, death, informed consent withdrawal, or study end, whichever comes first in combination with 1.3 mg/meter^2 (m^2) Bor administered subcutaneously (SC) once daily on Days 1, 4, 8 and 11 of each 21-day cycle along with 20 mg Dex via oral tablet or IV infusion once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for a total of 8 cycles.
- Daratumumab + Bor + Dex: Japanese participants with RRMM received 16 mg/kg Daratumumab IV infusion once weekly of each 21-day cycle in Cycle 1 to Cycle 3; once every 3 weeks on Day 1 of each 21-day cycle in Cycle 4 to Cycle 8; and once every 4 weeks on day 1 of each 28-day cycle from cycle 9 onwards until disease progression, intolerable toxicity, death, informed consent withdrawal, or study end, whichever comes first in combination with 1.3 mg/m^2 Bor administered SC once daily on Days 1, 4, 8 and 11 of each 21-day cycle along with 20 mg Dex oral tablet or IV infusion once daily on Days 1, 2, 4, 5, 8, 9, 11, and 12 of each 21-day cycle for a total of 8 cycles.
Period: Overall Study
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
Started | 10 | 14
Completed | 0 | 0
Not Completed | 10 | 14
Not completed — Death | 0 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ongoing | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 67.9 (11.02) | 70.9 (6.21) | 69.6 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 14 | 24
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as time from randomization until earliest date of disease progression (PD), determined by Independent Review Committee (IRC), according to the International Myeloma Working Group (IMWG) Response Criteria, or death due to any cause. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5 grams per deciliter {g/dL}]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200 milligrams per 24 hours {mg/24h}]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved serum free light chains (sFLC) levels [absolute increase >10mg/dL]; appearance of new lesion,>=50% increase from nadir in Sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: Up to approximately 32 months
Population: Intent-to-Treat (ITT) Population included all randomized participants whether or not randomized treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
Number analyzed (Participants) | 10 | 14
Months | NA [7.0 to NA] — The median and upper limit of 95% Confidence Interval were not estimable due to the length of follow-up in assessing the number of events. | 11.1 [4.9 to NA] — The upper limit of 95% Confidence Interval was not estimable due to the length of follow-up in assessing the number of events.
Statistical Analysis 1: Comparison: Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) vs Daratumumab + Bor + Dex; Test type: Other; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.11 to 1.52] — Hazard ratio was estimated using a Cox Proportional Hazards model stratified by the number of lines of prior therapy, prior bortezomib and revised international staging system (R-ISS) at screening, with a covariate of treatment

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from the date of randomization until the date of death due to any cause.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

3. Secondary Outcome: Duration of Response (DoR)
Description: DOR is defined as time from first documented evidence of partial response or better until first documented progression or death, whichever occurs first.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

4. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: Minimal Residual Disease (MRD) negativity rate is defined as the percentage of participants who are MRD negative by next generation sequencing (NGS).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

5. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as percentage of participants with a confirmed complete response (CR) or better (i.e., CR, stringent Complete Response (sCR)).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

6. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants with a confirmed partial response (PR) or better (i.e. PR, Very Good Partial Response [VGPR], CR or sCR).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

7. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR is defined as percentage of participants with a confirmed minimal response (MR) or better per International Myeloma Working Group (IMWG).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

8. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as time from the date of randomization and the first documented evidence of response (PR or better) among participants who achieve partial response or better.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

9. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization until the earliest date of documented PD or death due to PD. PD= increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5 grams per deciliter {g/dL}]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200 milligrams per 24 hours {mg/24h}]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved serum free light chains (sFLC) levels [absolute increase >10mg/dL]; appearance of new lesion,>=50% increase from nadir in Sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

10. Secondary Outcome: Progression-free Survival on Subsequent Line of Therapy (PFS2)
Description: PFS2 is defined as time from randomization to disease progression after initiation of new anti-myeloma therapy or death from any cause, whichever is earlier. If disease progression after new anti-myeloma therapy cannot be measured, a PFS event is defined as the date of discontinuation of new anti-myeloma therapy, or death from any cause, whichever is earlier
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA dictionary).
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Chemistry
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Urine Dipstick
Description: Urine samples will be collected for the urine dipstick analysis.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

15. Secondary Outcome: Number of Participants With Abnormal Ocular Findings on Ophthalmic Examination
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

16. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (Total Antibody)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

17. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (ADC)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

18. Secondary Outcome: Plasma Concentrations of Monomethyl Auristatin-F With a Cysteine Linker (Cys-mcMMAF)
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

19. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples will be collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

20. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples will be collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be further tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

21. Secondary Outcome: Number of Participants With Maximum Post-baseline Change From Baseline in Individual Items of Patient-reported Outcome Version of the Common Term Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a patient-reported outcome measure that was developed to evaluate symptomatic toxicities in patients in cancer clinical trials; it characterizes the frequency, severity, interference, and presence or absence of symptomatic toxicities. Responses ranges from 0 ("never," "none," "not at all," or "absent") to 4 ("almost constantly," "very severe," or "very much"), with a higher score indicating a higher frequency, severity, or interference of adverse events.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

22. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These included five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhoea, insomnia, dyspnoea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores are averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represent better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represent significant symptomatology. Baseline was defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

23. Secondary Outcome: Change From Baseline in HRQoL as Measured by EORTC IL52
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. For the EORTC IL52, disease symptoms domain of the QLQ-MY20 will be used for bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to100. A high score for disease symptoms represents a high level of symptomatology or problems.
Time Frame: Up to 255 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 32 months. The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Description: Safety population included all randomized participants who took at least 1 dose of study treatment.
Arm/Group | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) | Daratumumab + Bor + Dex
All-Cause Mortality (participants affected / at risk) | 0/10 | 4/14
Serious Adverse Events (participants affected / at risk) | 7/10 | 2/14
Other Adverse Events (participants affected / at risk) | 10/10 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) (N=10) | Daratumumab + Bor + Dex (N=14)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin + Bortezomib (Bor) + Dexamethasone (Dex) (N=10) | Daratumumab + Bor + Dex (N=14)
Malaise (General disorders) | 4 (4) | 3 (3)
Pyrexia (General disorders) | 2 (2) | 4 (5)
Injection site erythema (General disorders) | 3 (3) | 2 (2)
Sensation of foreign body (General disorders) | 3 (7) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (16) | 7 (14)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5)
Lymphopenia (Blood and lymphatic system disorders) | 2 (6) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (11) | 4 (6)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal erosion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (7) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Tinea cruris (Infections and infestations) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (6) | 5 (5)
White blood cell count decreased (Investigations) | 1 (1) | 4 (4)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 7 (13) | 0 (0)
Vision blurred (Eye disorders) | 7 (22) | 0 (0)
Dry eye (Eye disorders) | 3 (14) | 1 (1)
Eye irritation (Eye disorders) | 3 (8) | 1 (1)
Eye pain (Eye disorders) | 4 (10) | 0 (0)
Photophobia (Eye disorders) | 4 (16) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 2 (2)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Retinal haemorrhage (Eye disorders) | 2 (4) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0)
Conjunctival oedema (Eye disorders) | 1 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (4) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (2) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (6) | 4 (6)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (5)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (6)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (6) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT06868667/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT06868667/SAP_001.pdf